CLINICAL TRIAL: NCT04709900
Title: DYnamic CT Stress Myocardial perfusioN, CT Fractional Flow Reserve and Coronary CT Angiography for Optimized treatMent Strategy In Patients With sTable Chest Pain syndromEs
Brief Title: CT Stress Myocardial Perfusion, Fractional Flow Reserve and Angiography in Patients With Stable Chest Pain Syndromes
Acronym: DYNAMITE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Klaus Fuglsang Kofoed, Clinical associated Research Professor, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NNF19OC0057592
Record Dates: First submitted 2021-01-12; First posted 2021-01-14 (Actual); Last update posted 2022-12-12 (Actual); Status verified 2022-12

CONDITIONS: Coronary Artery Disease; Chest Syndrome; Acute Myocardial Infarction; Heart Failure; Stroke; Cardiovascular Diseases
Keywords: Cardiac CT; Chest pain; Coronary artery disease
MeSH Terms: conditions — Coronary Artery Disease; Heart Failure; Stroke; Cardiovascular Diseases; Chest Pain | interventions — Computed Tomography Angiography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Active Comparator): CT angiography, FFR-CT and dynamic CT stress myocardial perfusion guided treatment strategy
  Interventions: Diagnostic Test: CT angiography, FFR-CT and stress CT myocardial perfusion
- Standard care group (No Intervention): Evaluation and treatment strategy according to contemporary clinical practice

INTERVENTIONS:
Diagnostic Test: CT angiography, FFR-CT and stress CT myocardial perfusion — The study intervention team consists of a specialist in Cardiac CT imaging, an invasive cardiologist, a thoracic surgeon and a cardiology nurse specialist. Treatment strategy defined by the study team based on CT findings involve referral for percutaneous coronary intervention, Coronary Artery Bypass surgery and/or initiation of optimal medical therapy, in addition to potential supplementary diagnostic procedures.
  Arms: Intervention group

SUMMARY:
The purpose of the DYNAMITE trial (Dynamic CT stress myocardial perfusion, CT fractional flow reserve (FFR-CT) and coronary CT angiography for optimized treatment strategy in patients with chest pain syndromes) is to determine the ability of combined anatomical and functional cardiac CT imaging to improve morbidity and mortality in patients with suspected or known ischemic heart disease.

DETAILED DESCRIPTION:
Trial design

The DYNAMITE trial is an investigator-initiated, randomised controlled, open-labelled trial conducted in the Capital Region of Copenhagen, Denmark

The following hypothesis will be tested:

* First primary hypothesis: A treatment strategy guided by combined dynamic CT myocardial stress perfusion, FFR-CT and CT coronary angiography improves clinical outcome compared with a conventional management strategy in patients with chronic chest pain syndromes
* Second primary hypothesis: A treatment strategy guided by combined dynamic CT stress myocardial perfusion, FFR-CT and CT coronary angiography results in improved symptom relief compared with a conventional management strategy in patients with chronic chest pain syndromes

ELIGIBILITY:
Inclusion Criteria:

* Chest pain in patients with clinically suspected or confirmed ischemic heart disease
* Clinical indication for non-acute coronary evaluation
* Status of coronary revascularization

  1. With previous coronary revascularization - all patients
  2. Without previous coronary revascularization

     1. Age≥65 years - all patients with chest pain
     2. Age>50 - <65 years - typical angina pectoris and at least one cardiovascular risk factor and/or previous myocardial infarction

        * Typical angina requiring all 3 criteria present: a) constrictive discomfort in the front of the chest or in the neck, jaw, shoulder or arm, b) precipitated by physical exertion c) relieved by rest or nitrates within 5 min.
        * Cardiovascular risk factors: hypertension, diabetes, hypercholesterolemia, current smoking, family history of ischemic heart disease, previous stroke, peripheral artery disease

Exclusion Criteria:

* Persistent chest pain and signs of ongoing acute myocardial ischemia requiring acute coronary intervention
* Hospitalization and discharge with the confirmed diagnosis acute coronary syndrome (STEMI or NSTEMI) within the last 6 months
* Severe valvular heart disease as primary diagnosis and/or in potential need of percutaneous or surgical valve treatment
* Known severe heart failure (LVEF less than 35%)
* Language, cultural or mental factors preventing the patient from understanding the informed consent form
* Known atrial fibrillation
* Known renal impairment (estimated Glomerular Filtration Rate below <30 ml/min)
* Known x-ray contrast allergy
* Known intolerance to adenosine infusion

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2021-12-03 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2031-12 (Estimated)

PRIMARY OUTCOMES:
Major Adverse Cardiovascular Events | 3 years
  cardiovascular death, acute myocardial infarction, stroke or hospitalization for heart failure

SECONDARY OUTCOMES:
Individual components of the primary endpoint | 3 years
  cardiovascular death; acute myocardial infarction; stroke or hospitalization for heart failure
Acute myocardial infarction stratified by subtype | 12 months
  Subtypes of acute myocardial infarction according to Fourth Universal Definition 2018
Hospitalization due to unstable angina pectoris, bleeding, pacemaker and/or implantable/cardioverter defibrillator implantation, surgical or percutaneous heart valve treatment | 3 years
  Cardiovascular hospitalizations
All-cause mortality | 3 years
  All-cause mortality
All-cause mortality | 10 years
  Long-term registry based all-cause mortality at 10 years
Number and type of diagnostic tests performed | 12 months
  Cardiac CT, Exercise ECG, perfusion Positron Emission Tomography, perfusion Single-photon emission computed tomography, perfusion magnetic resonance, invasive coronary angiography, invasive fractional flow reserve, intravascular ultrasound, optical coherence tomography
Number of invasive coronary test not leading to coronary revascularization | 12 months
  number of invasive procedures
Number of coronary revascularization | 3 years
  Coronary bypass surgery and/or percutaneous coronary intervention
Cumulative iodinated contrast volume | 12 months
  Cardiac computed tomography, invasive coronary angiography, invasive fractional flow reserve, intravascular ultrasound, invasive optical coherence tomography
Cumulative radiation dose | 12 months
  Cardiac CT, perfusion Positron Emission Tomography, perfusion Single-photon emission computed tomography, perfusion magnetic resonance, invasive coronary angiography, invasive fractional flow reserve, intravascular ultrasound, optical coherence tomography
Major procedural complications occuring during procedures (invasive, non-invasive or coronary revascularization) | 12 months
  death, cardiac arrest, cardiac arrhytmia, acute myocardial infarction, stroke, bleeding, unplanned revascularization and any complication requiring and/or prolonging hospitalizaation at least 24 hours
Minor procedural complication specific to type of procedure (invasive, non-invasive or during coronary revascularization) | 12 months
  Minor procedural complications
Patients diagnosed with non-cardiac disease as likely explanation for symptoms | 12 months
  non-cardiac diseases causing chest pain
Seattle Angina Questionaire | 3 months and 12 months
  Seattle Angina Questionaire pre-randomization, 3 months and 12 months after randomization
Quality of life by EQ-5D-5L instrument | 3 months and 12 months
  Quality of life estimated by EQ-5D-5L instrument pre-randomization, 3 months and 12 months after randomization

CONTACTS AND LOCATIONS:
Overall Officials: Klaus F Kofoed, MD, Principal Investigator — Department of Cardiology, Rigshospitalet, University of Copenhagen, Denmark
Locations (1):
- Department of Cardiology and Radiology, Rigshospitalet, The Heart Center, Capital Region of Copenhagen, University of Copenhagen, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Following publication of the main results of the trial, anonymized data will be made available to other researchers through the Zenodo open data repository.
Supporting Information: Study Protocol, SAP
Time Frame: Statistical Analysis Plan and study protocol a time of publication
Access Criteria: Curated by principle investigator according to contemporary law